CLINICAL TRIAL: NCT04949295
Title: Evaluation of Ocular Surface in Hemodialysis Patients by Ocular Surface Analyzer
Status: Completed | Type: Observational
Sponsor: XiaoYong Liu (Other)
Responsible Party: Sponsor-Investigator, XiaoYong Liu, Deputy chief physician, First Affiliated Hospital of Jinan University
Organization: First Affiliated Hospital of Jinan University (Other)
Other Study IDs: 2021JN
Record Dates: First submitted 2021-06-26; First posted 2021-07-02 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Hemodialysis; Ocular Surface Disease; Dry Eye; OSDI
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the hemodialysis group: investigated with the OSDI scale, and then bilateral ocular surface examinations were performed with Keratograph5M eye surface comprehensive analyzer. Non-invasive tear meniscus height (NITMH), first tear film break-up time (FTBUT), average tear film break-up time (ATBUT), dry eye severity grade, tear film lipid layer analysis (distribution and color), tear film lipid layer thickness grade, meibomian gland opening blocking site, meibomian gland opening blocking analysis, meibomian gland opening secretion oil character score, eye redness index analysis (conjunctiva, ciliary shape), and meibomian gland absence area score were recorded.
  Interventions: Device: ocular surface analyzer
- the normal group: investigated with the OSDI scale, and then bilateral ocular surface examinations were performed with Keratograph5M eye surface comprehensive analyzer. Non-invasive tear meniscus height (NITMH), first tear film break-up time (FTBUT), average tear film break-up time (ATBUT), dry eye severity grade, tear film lipid layer analysis (distribution and color), tear film lipid layer thickness grade, meibomian gland opening blocking site, meibomian gland opening blocking analysis, meibomian gland opening secretion oil character score, eye redness index analysis (conjunctiva, ciliary shape), and meibomian gland absence area score were recorded.
  Interventions: Device: ocular surface analyzer

INTERVENTIONS:
Device: ocular surface analyzer — Using ocular surface analyzer for Inspection

SUMMARY:
We clinically observed that some hemodialysis patients had corneal epithelial dryness, shedding, edema, and persistent epithelial nonunion after ocular surgery, which seriously affected the effect of surgery, and it is necessary to study the ocular surface characteristics of hemodialysis patients. In this study, we examined the ocular surface and analyzed and investigated the characteristics of the ocular surface in hemodialysis patients to provide a basis for ocular surface intervention or treatment in hemodialysis patients before ocular surgery in clinical practice.

DETAILED DESCRIPTION:
This study is a clinical case-control study. A total of 36 hemodialysis patients and 36 normal subjects were randomly selected from the Nephrology Department of the First Affiliated Hospital of Jinan University .All the subjects in the hemodialysis group (n = 36, 72 eyes) and the normal group (n = 36, 72 eyes) were investigated with the OSDI scale, and then bilateral ocular surface examinations were performed with Keratograph5M eye surface comprehensive analyzer. Non-invasive tear meniscus height (NITMH), first tear film break-up time (FTBUT), average tear film break-up time (ATBUT), dry eye severity grade, tear film lipid layer analysis (distribution and color), tear film lipid layer thickness grade, meibomian gland opening blocking site, meibomian gland opening blocking analysis, meibomian gland opening secretion oil character score, eye redness index analysis (conjunctiva, ciliary shape), and meibomian gland absence area score were recorded.

ELIGIBILITY:
the hemodialysis group Inclusion Criteria:

* Older than 18
* Hemodialysis patient
* The subject understands the purpose of this clinical trial and agrees to sign an informed consent form.

the hemodialysis group Exclusion Criteria:

* Previous history of ocular trauma or surgery
* History of wearing contact lenses
* Can Not Stop the use of dry eye caused by drugs and other drugs may directly affect the stability of tear film tears
* Eyelid abnormalities (such as eyelid insufficiency, entropion and ECTROPION, tumor, severe trichiasis)
* There have been peritoneal dialysis, kidney transplant surgery patients.

the normal group Inclusion Criteria:

* Older than 18
* Healthy people do not have other systemic diseases, such as diabetes and hypertension
* The subject understands the purpose of this clinical trial and agrees to sign an informed consent form.

the normal group Exclusion Criteria:

* Previous history of ocular trauma or surgery
* History of wearing contact lenses
* Can Not Stop the use of dry eye caused by drugs and other drugs may directly affect the stability of tear film tears.

Ages: 25 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 36 hemodialysis patients and 36 normal subjects were randomly selected from the Nephrology Department of the First Affiliated Hospital of Jinan University .
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Non-invasive tear meniscus height | 1year
  Maximum and minimum of Non-invasive tear meniscus height in millimetre，higher scores mean a better outcome.
first tear film break-up time | 1year
  Maximum and minimum of first tear film break-up time in Seconds，higher scores mean a better outcome.
average tear film break-up time | 1year
  Maximum and minimum of average tear film break-up time in Seconds，higher scores mean a better outcome.
dry eye severity grade | 1year
  Maximum and minimum of dry eye severity grade，higher scores mean a worse outcome.
tear film lipid layer analysis (distribution and color) | 1year
  Maximum and minimum of tear film lipid layer analysis (distribution and color)，higher scores mean a better outcome.
tear film lipid layer thickness grade | 1year
  Maximum and minimum of tear film lipid layer thickness grade,higher scores mean a better outcome.
meibomian gland opening blocking site | 1year
  Maximum and minimum of meibomian gland opening blocking site，higher scores mean a worse outcome.
meibomian gland opening blocking analysis | 1year
  Maximum and minimum of meibomian gland opening blocking analysis，higher scores mean a worse outcome.
meibomian gland opening secretion oil character score | 1year
  Maximum and minimum of meibomian gland opening secretion oil character score，higher scores mean a worse outcome.
eye redness index analysis (conjunctiva, ciliary shape) | 1year
  Maximum and minimum of eye redness index analysis (conjunctiva, ciliary shape)，higher scores mean a worse outcome.
meibomian gland absence area score | 1year
  Maximum and minimum of meibomian gland absence area score，higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided